CLINICAL TRIAL: NCT02291783
Title: A Double-Blind, Placebo-Controlled, Single and Multiple Oral Dose, Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of HTL0009936 in Healthy Subjects
Brief Title: Phase I, Healthy Subject, Safety, Tolerability and Pharmacokinetic Study of an M1 Agonist to Treat Cognitive Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nxera Pharma UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9936-101; 2013-002307-34 (EudraCT Number)
Record Dates: First submitted 2014-10-07; First posted 2014-11-14 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HTL0009936 (Experimental): HTL0009936 single and multiple ascending oral doses.
  Interventions: Drug: HTL0009936
- HTL0009936 Placebo (Placebo Comparator): HTL0009936 matching placebo
  Interventions: Drug: HTL0009936 placebo

INTERVENTIONS:
Drug: HTL0009936 — Single dose
  Other Names: 9936, HTL0009936
  Arms: HTL0009936
Drug: HTL0009936 placebo — Placebo single dose
  Other Names: Placebo
  Arms: HTL0009936 Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics in young and elderly healthy volunteers of HTL9936, a selective M1 receptor agonist intended for the treatment of cognitive disorders.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics in young and elderly healthy volunteers of HTL9936, a selective M1 receptor agonist intended for the treatment of cognitive disorders. This study is a single ascending dose study.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of ≥19 and ≤ 30kg/m²
* Healthy subject free from any clinically significant illness or disease
* Female subjects must be ≥65 years

Exclusion Criteria:

* Subject who is predicted to be a CYP2D6 poor or ultra rapid metabolizer
* History of hypersensitivity to study drug
* History of epilepsy or seizures
* Subject with previous history of suicidal behavior
* Subjects with significant hearing impairment
* Subjects with an abnormal EEG

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events, as a measure of safety and tolerability | From signing of informed consent up to 30 days after the final visit
  AE reports include a description of the AE, date and time of onset and resolution, intensity, and relationship to IMP.
Changes in Safety Lab parameters as a measure of safety and tolerability | Screening, Day-1, at select dosing days, and at 5 to 7 days post dose for single doseand 15 to 17 days post first dose in multiple dosing.
  Hematology, clinical chemistry, urinalysis
Changes in vital signs as a measure of safety and tolerability | Screening, Day-1, at select dosing days and at 5 to 7 days post dose for single dose, and 15 to 17 days post first dose in multiple dosing.
  Pulse rate,body temperature,blood pressure, and orthostatic changes.
Changes in 12-lead electrocardiograms as a measure of safety and tolerability | Screening, pre-dose, at select dosing days and at 5 to 7 days post dose for single dose,and 15 to 17 days post first dose in multiple dosing.
  Change in ECG parameters

SECONDARY OUTCOMES:
Pharmacokinetic measures in plasma as measured by Peak plasma concentration (Cmax) | Pre-dose, multiple time points to 24h, at select dosing days, and 5 to 7 days post dosefor single dose,and 15 to 17 days post first dose in multiple dosing.
  Peak plasma concentration (Cmax), time at occurrence of Cmax (tmax), Area under the plasma concentration versus time curve (AUC) 0-t, 0- infinity, percent of AUC 0-infinity, Cmax normalized by dose, AUC 0-t normalized for dose.
Pharmacokinetic measures in cerebro spinal fluid (CSF) in young males as measured by max observed CSF (Cmax CSF) | Part 1 - 1h, 2h,3h post dose
  Maximum observed CSF concentration (Cmax CSF), area under the CSF concentration versus time
Pharmacokinetic measures to assess the food effect as measured by ANOVA | Pre-dose, multiple time points to 24h, and at 12h, 24h and 5 to 7 days post dose.
  Food effect analysis will be based on analysis of variance (ANOVA) for treatment differences.
Pharmacodynamic response as measured by pupillometry | Multiple time points Day1 to 6h post dose Part 1 only.
  Changes in average pupil diameter as measured in 3 different conditions of lux.
Pharmacokinetic measures in urine in young males and elderly male and female subjects as measured by amount of urine excreted at collection intervals | Pre-dose,multiple 4h collection intervals to 24h post dose on select dosing days to Day 10 for multiple dosing.
  Amount excreted in urine at each collection interval (Ae1-t2) all parts. Cumulative amount excreted to 12h and 24h (Ae0-t) depending on Part. Cumulative urine excreted of unchanged drug to 24h (Fe%) and to 12h depending on Part. Volume of urine collected during each collection interval (Vur), and renal clearance (CLr) all parts
Pharmacodynamic response as measured by Bond and Lader visual analogue scale | Day 1 at multiple timepoints to 24h post dose.
  Changes in 3 factor scores (Alertness, Contentedness and Calmness) which will be derived from the individual VAS scores
Pharmacodynamic response as measured by changes in qEEG and Event Related Potentials (ERP) | Screening, Day-1, Day 4, Day 9 multiple dosing regimen only
  qEEg and ERP (P50 sensory gating, Mismatch Negativity and P300)

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, MBChB, Principal Investigator — Parexel
Locations (1):
- Parexel Early Phase Clinical Unit, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No